CLINICAL TRIAL: NCT06132906
Title: Comparison of Accuracy Between Novel Locating Guide Design With Pre-bent Titanium Plates and 3d Printed Intermediate Wafer to Reposition the Maxilla After le Fort 1 Osteotomy in Orthognathic Surgery
Brief Title: Comparison Between Two Techniques to Reposition the Maxilla After le Fort 1
Acronym: orthognathic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: orthognathicalexu
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Dentofacial Deformities; Le Fort; I
Keywords: orthognathic; virtual planning
MeSH Terms: conditions — Dentofacial Deformities | interventions — Orthognathic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Study group) will be treated with locating guides to reposition the maxilla with pre-bent plates (Experimental): After le fort 1 osteotomy, locating guides will be used to reposition the maxilla with pre-bent plates.
  Interventions: Procedure: Orthognathic surgery (lefort1)
- (Control group) will be treated with Intermediate wafer. (Active Comparator): After le fort 1 osteotomy, Intermediate wafer will be used with intermaxillary fixation.
  Interventions: Procedure: Orthognathic surgery (lefort1)

INTERVENTIONS:
Procedure: Orthognathic surgery (lefort1) — 1. All patients will be treated under general anesthesia.
  2. The surgical field will be scrubbed with povidone-iodine surgical scrub solution, followed by draping of the patient with sterile towels exposing only the area of surgery.
  3. The surgical procedure of Le Fort I osteotomy will be performed which can be summarized as follows:
     1. External reference marking
     2. Incision and subperiosteal dissection
     3. Maxillary osteotomy
     4. Pterygomaxillary disjunction,
     5. Septal, vomerine, and lateral nasal osteotomies
     6. Down fracture
     7. Mobilization of the maxilla
     8. Application of stent in one group and the locating guide in the other group.
     9. Maxillary fixation
     10. Occlusal evaluation
     11. Wound debridement and closure

SUMMARY:
clinical and radiographic comparison between novel locating guide design with pre-bent titanium plates and 3d printed intermediate wafer to reposition the maxilla after Le Fort 1 osteotomy in orthognathic surgery (randomized controlled clinical trial)

DETAILED DESCRIPTION:
Eligible patients will be allocated randomly into 2 equal groups with 7 patients in each group according to the method that will be used to reposition the maxilla by simple randomization using computer generated random numbers. Group 1 (Study group) will be treated with locating guides to reposition the maxilla with pre-bent plates on 3d model. Group 2 (Control group) will be treated with Intermediate wafer.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring Le Fort I osteotomy will be selected including those suffering from skeletal malocclusion (Class II or Class III), midface hypoplasia or vertical maxillary excess.

Exclusion Criteria:

cleft lip and palate. skeletal disharmony due to trauma or severe facial asymmetry. significant medical condition.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation of accuracy by superimposition | 2 weeks
  Postoperative CBCT was obtained after 2 weeks of surgery for comparison with the expected position of the maxilla in the preoperative virtual plan using 3-matic software in Mimics innovation suite software package. The preoperative planned final maxillary position was compared with the actual postoperative maxillary position by superimposing both STL models on each other with anatomical points along the orbital rims and the zygomatic arch used as reference points for alignment. The N points registration tool was used to obtain the alignment. Afterwards, using trim tool all parts were trimmed except that between the plates and the maxillary teeth crowns. Then the part comparison analysis tool was used to calculate the accuracy of the superimposition of the maxillary segment using point-based analysis algorithm after 2 weeks of surgery for comparison with the expected position of the maxilla in the preoperative virtual plan using Mimics innovation suite software.
The surgery duration | 1 week
  The time taken between performing the Le fort 1 osteotomy till completion of plate fixation will be measured.

SECONDARY OUTCOMES:
Postoperative Pain | after one week, two weeks
  Will be assessed through a 10-point Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Faculty of dentistry, Alexandria, Egypt